CLINICAL TRIAL: NCT06449755
Title: Elastic Nail Versus Screw for Closed Reduction and Intramedullary Fixation of Displaced Fractures of the Fifth Metacarpal Neck: a Randomised Controlled Trial
Brief Title: Elastic Nail Versus Screw for Intramedullary Fixation of Displaced Fractures of the Fifth Metacarpal Neck
Acronym: Boxerfx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, AHMET MUCTEBA YILDIRIM, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 159108493
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Metacarpal Fracture; Boxer's Fracture
MeSH Terms: interventions — Diagnostic Imaging; Hand Strength

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elastic Nail (Other): Percutaneous antegrade elastic nail fixation
  Interventions: Diagnostic Test: Radiologic examination; Procedure: Grip Strength; Other: Quick DASH Questionnaire
- Screw (Other): Percutaneous retrograde screw fixation
  Interventions: Diagnostic Test: Radiologic examination; Procedure: Grip Strength; Other: Quick DASH Questionnaire

INTERVENTIONS:
Diagnostic Test: Radiologic examination — Posoperative first week, month and third month On the x-ray of Hand AP view: metacarpal shortening On the x-ray of Hand 30 degree pronation view: dorsal angulation
Procedure: Grip Strength — Postoperative first month and third month grip streng compare with Cambry hand dinamometer.
Other: Quick DASH Questionnaire — Quick DASH is an 11-question questionnaire that assesses upper extremity functionality.

SUMMARY:
The goal of this clinical trial is to compare two different intramedullary fixation technique in patient diagnosed with deplased fifth metacarpal neck fracture. The main questions it aims to answer are:

* Can percutaneous screw application be a more stable fixation method than intramedullary elastic nail application?
* Can screw application create a significant difference in the recovery of grip strength in the early period compared to elastic nail application? Patients will be followed up at the 1st week, 1st month and 3rd month postoperatively. Functionality will be evaluated with Quick DASH score at the 3rd month. At the 1st and 3rd month controls, grip strength will be evaluated. At the same time, metacarpal shortening and angulations will be measured on x-ray. Researchers will compare percutaneous screw and elastic nail group to see grip strength, healing time and radiologic parameter difference.

DETAILED DESCRIPTION:
In this study, patients admitted to the emergency department with displaced fifth metacarpal neck fracture will be included. Exclusion criteria will include patients with other concomitant trauma, open fractures, fractures with intraarticular joint extension, and previous hand surgery in which the hand anatomy was distorted. Patients between the ages of 18 and 60 who have more than 30 degrees of angulation from the 30 degree hand pronation radiograph at admission and who consent to surgery will be included in the study. One of the two groups in the study will undergo closed reduction followed by percutaneous intramedullary retrograde screw fixation, while the other group will undergo intramedullary antegrade elastic nail application. Patients will be followed up with ulnar gutter splint for the first week postoperatively. After the first week, the splint will be removed and range of motion, gripping and pinching exercises will be given to the patients.

Radiological examinations (dorsal angulation and metacarpal shortening will be measured) will be performed in the first week, first and third months postoperatively. Hand grip strength will be measured with Cambry dynamometer at the first and third month. At the 3rd month, upper extremity functionality will be evaluated with Quick DASH score and a comparison will be made between the two groups.

Randomisation will be performed with an internet-based application. Clinical ethics committee approval was obtained before the study started.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-60 years with displaced fifth metacarpal fractures with angulation greater than 30 degrees

Exclusion Criteria:

* Open fracture
* Patients with multiple injuries
* History of hand surgery
* Intraarticular metacarpal neck fractures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Dorsal Angulation and Metacarpal Shortening | Preoperative, Postoperative first week, first and third month
  Measurement of dorsal angulation between two fracture fragments on a hand oblique 30-degree pronation X-Ray Measurement of shortness of the fifth metacarpal on hand AP X-ray

SECONDARY OUTCOMES:
Grip Strength | Postoperative first and third month
  Hand grip strength will be measured with CAMBRY hand dynamometer at 1 and 3 months postoperatively.

OTHER OUTCOMES:
Healing Time | Preoperative, Postoperative first week, first and third month
  In follow-up X-rays, complete osseous bridging in 3 of 4 cortices and absence of pain in the patient will be taken as a sign of healing.
Upper Extremity Functionality | Postoperative third month
  Patients will be evaluated at the 3rd postoperative month with the Quick DASH 11-question questionnaire assessing upper extremity functionality.

CONTACTS AND LOCATIONS:
Overall Officials: Serkan MD Bayram, MD, Principal Investigator — Assistant Professor
Locations (1):
- Istanbul Unıversity Medicine Faculty Orthopaedic Department, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No